CLINICAL TRIAL: NCT04985656
Title: A Phase 2, Open-Label Study of Intravenous Pevonedistat in Combination With Oral Decitabine and Cedazuridine in Adult Patients With Higher-Risk Myelodysplastic Syndromes
Brief Title: A Study of Pevonedistat Combined With Decitabine and Cedazuridine in Adults With Higher-risk Myelodysplastic Syndromes
Acronym: PEVOBINE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision to Terminate Trial
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pevonedistat-2003
Record Dates: First submitted 2021-07-29; First posted 2021-08-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Drug Therapy
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — pevonedistat; Decitabine; cedazuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pevonedistat 20 mg/m^2 + Decitabine 35 mg + Cedazuridine 100 mg (Experimental): Pevonedistat 20 mg/m^2, 60-minute intravenous (IV) infusion, once daily, on Days 1, 3, and 5 in each 28-day cycle in combination with decitabine 35 mg and cedazuridine 100 mg tablets, orally, once daily on Days 1 through 5 in each 28-day cycle up to 30 months.
  Interventions: Drug: Pevonedistat; Drug: Decitabine; Drug: Cedazuridine

INTERVENTIONS:
Drug: Pevonedistat — Pevonedistat IV infusion
Drug: Decitabine — Decitabine tablets
Drug: Cedazuridine — Cedazuridine tablets

SUMMARY:
The main aim of the study is to see if signs and symptoms of myelodysplastic syndromes disappear when treated with pevonedistat combined with decitabine and cedazuridine.

Participants will receive an infusion of pevonedistat 3 times during a 28-day cycle. They will also take decitabine and cedazuridine tablets once a day for the first 5 days of the same cycle. A minimum of 6 28-day cycles is recommended, but participants can stop treatment at any time.

A bone marrow biopsy, bone marrow aspirates, and blood samples will be collected during the study.

Participants will attend a follow-up visit 30 days after their last dose of pevonedistat. Once treatment has ended, participants will be followed up with either monthly clinic visits or will be contacted every 3 months.

DETAILED DESCRIPTION:
The drug being tested in this study is called Pevonedistat (TAK-924/MLN4924). Pevonedistat is being tested to treat people who have higher-risk myelodysplastic syndromes (HR MDS). This study will look at the overall survival, event free survival and response in people who take pevonedistat in combination with oral decitabine and cedazuridine in addition to standard care.

The study will enroll approximately 94 patients. Participants will be assigned to following treatment group:

• Pevonedistat 20 mg/m^2 + Decitabine 35 mg + Cedazuridine 100 mg

All participants will receive pevonedistat in combination with decitabine and cedazuridine as specified in the protocol.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is approximately 30 months. Participants will make multiple visits to the clinic and will be contacted by telephone OR plus a final visit after receiving their last dose of drug/compound 30 days after last dose of study drug for event free survival (EFS) follow-up followed by overall survival (OS) follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Documented morphologically confirmed diagnosis of HR MDS according to the 2016 World Health Organisation (WHO) classification.
2. All participants must also have one of the following Prognostic Risk Categories based on the Revised International Prognostic Staging System (IPSS-R): Very high >6 points, high (4.5 to 6 points), or intermediate >3 to 4.5 points. Participants in the intermediate category must have >5% bone marrow myeloblasts.
3. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of ≤2.
4. Able to undergo the study-required bone marrow sample collection procedures.
5. Suitable venous access for the study-required blood sampling (i.e., including pharmacokinetic (PK) sampling).
6. Known Human Immunodeficiency Virus (HIV)-positive participants who meet the following criteria will be considered eligible:

   * Cluster of differentiation 4 (CD4) count >350 cells per cubic millimeter (cells/mm^3).
   * Undetectable viral load.
   * Maintained on modern therapeutic regimens.
   * No history of Acquired Immune Deficiency Syndrome (AIDS)-defining opportunistic infections.

Exclusion Criteria:

1. Histologically or cytologically documented diagnosis of Acute Myelogenous Leukemia (AML) or Chronic Myelomonocytic Leukemia (CMML).
2. Previous treatment for HR MDS with chemotherapy or other antineoplastic agents, including hypomethylating agents (HMAs), such as decitabine or azacitidine. Previous treatment is permitted with hydroxyurea and with lenalidomide, except that lenalidomide may not be given within 8 weeks before the first dose of study drug(s).
3. Have known hypersensitivity to pevonedistat or its excipients.
4. Have known hypersensitivity to oral decitabine and cedazuridine or its excipients.
5. Diagnosed or treated for another malignancy within 2 years before enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.
6. Participants with either clinical evidence of or history of central nervous system (CNS) involvement.
7. Are known hepatitis B surface antigen seropositive, or known or suspected active hepatitis C infection. (Note: Participants who have isolated positive hepatitis B core antibody [i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody] must have an undetectable hepatitis B viral load. Participants with history of hepatitis C virus [HCV] infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.)
8. Have known hepatic cirrhosis or severe pre-existing hepatic impairment.
9. Have known cardiopulmonary disease, defined as unstable angina, clinically significant arrhythmia, congestive heart failure (New York Heart Association Class III or IV), and/or myocardial infarction within 6 months before first dose, or severe pulmonary hypertension. As an example, well-controlled atrial fibrillation (AF) would not be an exclusion, whereas uncontrolled AF would be an exclusion.
10. Have positive test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection that is laboratory confirmed by a reverse transcription polymerase chain reaction (RT-PCR) test at screening. Testing related to coronavirus disease 2019 (COVID-19) must be performed according to institutional policy and/or per local regulatory guidelines.
11. Participants who have had a known infection of SARS-CoV-2 or COVID-19 are permitted if COVID-19 RT-PCR test is negative prior to the screening visit and they present with no symptoms. Participants with documented vaccination history for COVID-19 do not need to be tested, unless they are symptomatic, according to institutional policy and/or local regulatory guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-01-08 (Estimated); Study Completion 2024-11-08 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) Rate | Up to 30 months
  CR Rate is defined as percentage of participants with HR MDS who achieve CR. CR for HR MDS as per the Modified IWG Response Criteria is defined as ≤5% myeloblasts with normal maturation of all cell lines in the bone marrow, and ≥11 grams per deciliter (g/dL) Hemoglobin (Hb), ≥100*10^9 per liter (/L) platelets (pl), ≥1.0*10^9/L neutrophils and 0% blasts in peripheral blood.

SECONDARY OUTCOMES:
Duration of Complete Remission (DOR) | Up to 30 months
  DOR is defined as the time that criteria are met for CR to the date of first documented disease progression or relapse after CR for responders of CR. CR for HR MDS as per modified IWG response criteria is defined as ≤5% myeloblasts with normal maturation of all cell lines in the bone marrow, and greater than or equal to (≥)11 g/dL hemoglobin (Hgb), ≥100*10^9/liter (/L) platelets (pl), ≥1.0*10^9/L neutrophils and 0% blasts in peripheral blood.
Overall Response Rate (ORR) | Up to 30 months
  ORR as per the modified IWG criteria for MDS is defined as percentage of participants with CR or partial remission (PR), CR: ≤5% myeloblasts with normal maturation of bone marrow (BM) cell lines, ≥11g/dL Hb, ≥100*10^9/L platelets, ≥1.0*10^9/L absolute neutrophil count (ANC), 0% blasts in peripheral blood. PR: all CR criteria met except bone marrow blasts ≥50% decrease over pretreatment but still >5%.
Time to First CR or PR or Hematologic Improvement (HI) | Up to 30 months
  It is defined as the time from the date of first dose of combination treatment to the first documented CR or PR or HI. CR: ≤5% myeloblasts with normal maturation of all bone marrow cell lines, ≥11 g/dL Hb, ≥100*10^9/L platelet, ≥1.0*10^9/L ANC, 0% blasts in peripheral blood; PR: all CR criteria met except bone marrow blasts ≥50% decrease over pretreatment but still >5%. HI: Hb increase ≥1.5 g/dL if pretreatment <11 g/dL; platelets absolute increase ≥30*10^9/L if baseline>20*10^9/L or increase from <20*10^9/L to >20*10^9/L and by at least 100%; neutrophil increase by 100% and absolute increase of >0.5*10^9/L if baseline <1.0*10^9/L.
Percentage of Participants with Hematologic Improvement | Up to 30 months
  HI for HR MDS is defined as per Modified IWG Response Criteria for MDS. HI: Hb increase ≥1.5 g/dL if pretreatment <11 g/dL; platelets absolute increase ≥30*10^9/L if baseline>20*10^9/L or increase from <20*10^9/L to >20*10^9/L and by at least 100%; neutrophil increase by 100% and absolute increase of >0.5*10^9/L if baseline <1.0*10^9/L.
Percentage of Participants with Red Blood Cell (RBC) Transfusion Independence, Platelet Transfusion Independence, and RBC and Platelet Transfusion Independence | Up to 30 months
  A participant is defined as RBC and/or platelet transfusion-independent if they receive no RBC and/or platelet transfusions for a period of at least 8 weeks during the time-period from the first dose of study drug administration through 30 days after the last dose of any study drug. Rate of RBC and/or platelet transfusion independence is defined as the percentage of participants who become RBC and/or platelet transfusion-independent divided by the number of participants who are RBC and/or platelet transfusion-dependent at Baseline.
Duration of RBC Transfusion Independence, Platelet Transfusion Independence, and RBC and Platelet Transfusion Independence | Up to 30 months
  The duration of transfusion independence is defined as the longest time between the last RBC and/or platelet transfusion before the start of the RBC and/or platelet transfusion-independent period and the first RBC and/or platelet transfusion after the start of the transfusion-independent period, which occurs at least 8 weeks later.
Overall Survival (OS) | Up to 30 months
  OS is defined as the time from the date of first dose of combination treatment to the date of death due to any cause.
Event Free Survival (EFS) | Up to 30 months
  EFS is defined as the time from the date of first dose of combination treatment to the date of the occurrence of an EFS event. An EFS event is defined as death or transformation to acute myelogenous leukemia (AML), whichever occurs first.
Plasma Concentration-Time Profile for Pevonedistat and Oral Decitabine and Cedazuridine | Days 1, 3 and 5 of each cycle pre-dose and at multiple time points (up to 30 months) post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/610983f7beb21d002a9260bb